CLINICAL TRIAL: NCT03494413
Title: Evaluation of Transpharyngeal Doppler Sonography as a Cerebral Monitoring Tool in Cardiac Surgery
Brief Title: Transpharyngeal Doppler Sonography for Cerebral Perfusion Monitoring
Acronym: TaPaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-00566
Record Dates: First submitted 2018-04-03; First posted 2018-04-11 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Cerebral Perfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 patients (1-20) validation arm (Experimental): Accuracy of cerebral flow measurement between TPS and CDS in 20 patients undergoing cardiovascular surgery with cardiopulmonary bypass
  Interventions: Diagnostic Test: Transpharyngeal Doppler sonography (TPS); Diagnostic Test: Conventional colour-coded Duplex sonography (CDS)
- 20 patients (21-40) HCA arm (Experimental): Assessment and comparison of TPS and CDS in hypothermic circulatory arrest (HCA) during cardiovascular surgery
  Interventions: Diagnostic Test: Transpharyngeal Doppler sonography (TPS); Diagnostic Test: Conventional colour-coded Duplex sonography (CDS)

INTERVENTIONS:
Diagnostic Test: Transpharyngeal Doppler sonography (TPS) — Usage of transpharyngeal Doppler to assess cerebral perfusion during cardiovascular surgery
Diagnostic Test: Conventional colour-coded Duplex sonography (CDS) — Usage of conventional colour-coded Duplex sonography (CDS) to assess cerebral perfusion during cardiovascular surgery

SUMMARY:
This prospective interventional study investigates transpharyngeal sonography (TPS) as an additional neuromonitoring strategy to assess cerebral perfusion during cardiovascular surgery. In the first part of the study the investigators will investigate the feasibility of TPS for visualization of aortic arch branches including the innominate and the carotid arteries in patients undergoing cardiac surgery with cardiopulmonary bypass. In the second part the investigators plan to adopt the investigators previous experiences on TPS to a selected population of patients undergoing ascending aortic and/or arch repair in hypothermic circulatory arrest (HCA).

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular Surgery
* Age > 18 yrs
* Informed Consent

Exclusion Criteria:

* Contraindication for TPS
* Carotid artery stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of cerebral flow velocity measurement | intraoperative phase, expected to be ca. 4 hours
  Cerebral blood flow velocity measurements will be performed with transpharyngeal Doppler sonography (TPS) and conventional colour-coded Duplex sonography (CDS). Doppler flow velocities (obtained at the same intraoperative phase and at the same time) will be compared between TPS and CDS TPS and different Doppler techniques.

SECONDARY OUTCOMES:
Hypothermic Circulatory Arrest | intraoperative phase, expected to be ca. 4 hours
  Doppler flow velocities (obtained with both methods in the Phase of hypothermic circulatory arrest - intraoperatively) will be compared between TPS and CDS TPS and different Doppler techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Inselspital, University Hospital Bern, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No